CLINICAL TRIAL: NCT05540249
Title: Effects of Pre-operative Oral Carbohydrates on Insulin Resistance and Postoperative Recovery in Diabetic Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Pre-operative Carbohydrates in Diabetic Patients Undergoing CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Wei Feng, Clinical Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-ZX40
Record Dates: First submitted 2022-09-03; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Insulin Resistance; Diabetes Mellitus, Type 2; Coronary Artery Bypass Surgery
Keywords: preoperative carbohydrates; diabetes mellitus; off-pump coronary artery bypass grafting; insulin resistance
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeons, anesthesiologists, ICU staff, nurses, outcome assessors, data collectors and data analysts will be blinded to the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CHO (Experimental): Patients in Group CHO will orally consume CHO 355ml containing 50 g of carbohydrates 8-12 hours before operation (20:00 -24:00 the evening before operation).
  Interventions: Dietary Supplement: carbohydrates
- Group CTRL (No Intervention): Patients in Group CTRL will consume no food or drink 12 hours before operation (20:00 the evening before operation).

INTERVENTIONS:
Dietary Supplement: carbohydrates — Patients will orally consume 355mL CHO after 20:00 the evening before surgery.
  Other Names: Outfast
  Arms: Group CHO

SUMMARY:
Preoperative carbohydrates (CHO) supplement has been shown to alleviate postoperative insulin resistance (IR) in nondiabetic patients undergoing a variety of surgeries. However, it remains controversial whether preoperative CHO could yield similar effects in diabetic patients. Thus, the investigators design a randomized controlled trial investigating the impact of preoperative CHO on postoperative IR and clinical outcomes in diabetic patients undergoing cardiac surgery. The results of the study may give some clinical implications and further improve perioperative care for diabetic patients.

DETAILED DESCRIPTION:
CHO supplement has been widely investigated in nondiabetic patients undergoing various surgeries. It has been proved that preoperative CHO could alleviate postoperative insulin resistance (IR) and improve patients' well-being in nondiabetic patients. However, whether preoperative CHO could yield similar effects in diabetic patients remains controversial. Till now, seldom has the administration of preoperative CHO been investigated in diabetic patients and few studies reported IR and postoperative recovery of diabetic patients undergoing cardiac surgery. The investigators present a prospective, single-center, single-blind, randomized, no-treatment controlled trial of preoperative CHO on diabetic patients undergoing off-pump coronary artery bypass grafting (OPCAB). A total of 62 patients will be enrolled and randomized to either Group CHO or Group control (CTRL). Patients in group CHO will receive CHO fluid containing 50 g of carbohydrates the evening before surgery (20:00-24:00) while their counterparts in Group CTRL will be fasted after 20:00 the evening before surgery. The primary endpoints are postoperative insulin resistance (IR) assessed via homeostasis model assessment (HOMA). The secondary endpoints are the potential mediators relating to IR including inflammatory factors and stress reactions assessed by serum cortisol. Exploratory endpoints are in-hospital clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed T2DM
2. Diagnosed with CAD with coronary angiography and indicated for OPCAB
3. Age between 18 and 75 years old
4. First operation in the morning and anesthesia induced around 8:00
5. Written informed consent by the patients

Exclusion Criteria:

1. Combined with other heart diseases or vascular malformations that require surgery in addition to OPCAB
2. Presence of symptoms or signs of heart failure such as orthopnea, distended jugular vein, lower extremity edema, etc.
3. Reduced LVEF (lower than 50%)
4. Combined with gastroesophageal reflux
5. Combined with thyroid insufficiency requiring replacement therapy with levothyroxine
6. Combined with adrenal insufficiency requiring replacement therapy with corticosteroids
7. Refuse to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Peri-operative Change from baseline HOMA-IR | Before anesthesia induction
  HOMA-IR = [blood insulin (mu/L) × Blood glucose (mmol/L)]/22.5
Peri-operative Change from baseline HOMA-IR | Immediately after surgery
  HOMA-IR = [blood insulin (mu/L) × Blood glucose (mmol/L)]/22.5
Peri-operative Change from baseline HOMA-IR | The first morning after surgery
  HOMA-IR = [blood insulin (mu/L) × Blood glucose (mmol/L)]/22.5
Peri-operative Change from baseline HOMA-IR | The second morning after surgery
  HOMA-IR = [blood insulin (mu/L) × Blood glucose (mmol/L)]/22.5
Peri-operative Change from baseline HOMA-IR | The third morning after surgery
  HOMA-IR = [blood insulin (mu/L) × Blood glucose (mmol/L)]/22.5
Peri-operative Change from baseline HOMA-IR | The fifth morning after surgery
  HOMA-IR = [blood insulin (mu/L) × Blood glucose (mmol/L)]/22.5

SECONDARY OUTCOMES:
Interleukin -1 (IL-1) | The first morning after surgery
  Inflammatory factors
Interleukin-6 (IL-6) | The first morning after surgery
  Inflammatory factors
Interleukin-8 (IL-8), | The first morning after surgery
  Inflammatory factors
Interleukin-10 (IL-10), | The first morning after surgery
  Inflammatory factors
Tumor necrosis fator-α (TNF-α) | The first morning after surgery
  Inflammatory factors
High-sensitivity C-reactive protein (hs-CRP) | The first morning after surgery
  Inflammatory factors

OTHER OUTCOMES:
Nausea or vomiting | In-hospital period after surgery (up to day 5)
  Nausea or vomiting requiring medical treatment such as ondansetron
New-onset postoperative atrial fibrillation (POAF) | In-hospital period after surgery (up to day 5)
  POAF is defined as new onset atrial fibrillation lasting at least 10min on the electrocardiogram (ECG) monitor or atrial fibrillation that requires treatment with medication after surgery.
Major adverse cardiovascular and cerebral events (MACCEs) | In-hospital period after surgery (up to day 5)
  A composite endpoints of all-cause death, non-fatal myocardial infarction, stroke.
ICU length | In-hospital period after surgery (up to day 5)
  The length of patient's stay in the ICU
Mechanical ventilation time | In-hospital period after surgery (up to day 5)
  Duration of patient ventilator-assisted breathing

IPD SHARING:
Plan to Share IPD: Yes
Except for the identifying data such as patients name and admission ID, all the IPD could be available to other researchers on reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: The data will become available after the publication of the study report.
Access Criteria: IPD could be accessed on reasonable request after approval of the principal investigator.